CLINICAL TRIAL: NCT02862951
Title: Sleep Efficiency and Quantification After Labor Epidural Analgesia
Acronym: Actiwatch
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Mohamed Tiouririne, MD, Anesthesiology attending, University of Virginia
Other Study IDs: 18682
Record Dates: First submitted 2016-06-16; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-08

CONDITIONS: Pregnancy
Keywords: pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Term pregnancy (>37 weeks gestation): Term pregnancy (>37 weeks gestation)

SUMMARY:
The specific aim is to attempt to quantify the amount and efficiency of sleep that parturients receive after placement of labor epidural analgesia.

DETAILED DESCRIPTION:
The hypothesis is that the placement of labor epidural analgesia results in improved sleep efficiency and increased amount of sleep for parturients during their labor process as measured by an actigraph. An actigraph is a watch that monitors movement and allows for non-invasive determination of sleep-wake cycles. For this study, the Actiwatch 2 will be used due to departmental availability. For this study, 36 parturients will be enrolled that are coming in for induction of labor at term gestational age, regardless of whether they think they will desire epidural analgesia or not . These parturients will wear the Actiwatch from the beginning of induction of their labor until the delivery of their baby. Participants will be instructed to press a button on the watch to record the start and end times of when they are trying to sleep. The data will then be analyzed to determine the amount of time that participants were able to sleep after placement of an epidural catheter as well as their sleep efficiency, defined as the percentage of time spent sleeping during the time in which sleep is attempted.

ELIGIBILITY:
Inclusion Criteria:

* Parturients admitted for induction of labor
* Term pregnancy (>37 weeks gestational age)

Exclusion Criteria:

* Preterm pregnancy (< 37 weeks gestational age) Parturients not willing or not able to give informed consent Patients receiving magnesium treatment will be excluded.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Parturients admitted for induction of labor
  -Term pregnancy (>37 weeks gestational age)
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
amount of sleep as measured by actiwatch device in hours of sleep | after placement of epidural analgesia until delivery
  Amount of sleep that parturients receive after placement of labor epidural analgesia.

SECONDARY OUTCOMES:
efficacy of sleep, automatically derived from the actiwatch device as restlessness during sleep | after placement of epidural analgesia until delivery
  Sleep efficiency is defined as the percentage of time spent sleeping during the time in which sleep is attempted.

CONTACTS AND LOCATIONS:
Overall Officials: Tiouririne Mohamed, MD, Principal Investigator — University of Virginia Dept of Anesthesiology
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Skowronski GA. Pain relief in childbirth: changing historical and feminist perspectives. Anaesth Intensive Care. 2015 Jul;43 Suppl:25-8. doi: 10.1177/0310057X150430S106. PMID 26126073
- [Background] Hall WA, Stoll K, Hutton EK, Brown H. A prospective study of effects of psychological factors and sleep on obstetric interventions, mode of birth, and neonatal outcomes among low-risk British Columbian women. BMC Pregnancy Childbirth. 2012 Aug 3;12:78. doi: 10.1186/1471-2393-12-78. PMID 22862846
- [Background] Wangel AM, Molin J, Ostman M, Jernstrom H. Emergency cesarean sections can be predicted by markers for stress, worry and sleep disturbances in first-time mothers. Acta Obstet Gynecol Scand. 2011 Mar;90(3):238-44. doi: 10.1111/j.1600-0412.2010.01056.x. Epub 2011 Feb 3. PMID 21306317